CLINICAL TRIAL: NCT05390957
Title: A Pilot Study of a Revised Online Chronic Pain Treatment for Military, RCMP, and Veterans
Brief Title: Pilot Study of Revised Online Chronic Pain Treatment for Military and Veterans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Pamela L. Holens, Principal Investigator, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS25212 (H2021:368)
Record Dates: First submitted 2022-01-08; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: The study is an open label, single site, single arm, pilot study. The primary goal of the study is to examine the efficacy of the ABBT-R program via comparison of pre-treatment and post-treatment scores on measures of pain and other related concerns, as well as examination of participant satisfaction with the program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): All participants in this pilot study will complete the active treatment
  Interventions: Behavioral: Acceptance Based Behavioural Therapy - Revised

INTERVENTIONS:
Behavioral: Acceptance Based Behavioural Therapy - Revised — The study intervention is a revised, updated version of a previously studied eight-module (8-week) online, acceptance-based behavioural therapy (ABBT) for chronic pain that was tailored specifically to a military, RCMP, and veteran population. The online treatment material is administered via the WebCAPSI Therapy program.

SUMMARY:
This study is being conducted to examine the efficacy of a revised version of an online chronic pain intervention tailored specifically for military, RCMP, and veterans. The original intervention from which the revised version emanates is an online psychotherapy for chronic pain that was developed using materials derived from cognitive behavioural therapy (CBT) and acceptance and commitment therapy (ACT) and has thus been described as an acceptance-based behavioural therapy (ABBT). For the purposes of this study, the revised intervention will be known as ABBT-R. The revised treatment protocol was developed based on feedback from participants who had engaged with the original version of the treatment protocol and who participated in a focus group study about their experiences with the intervention. It is hoped that the revised treatment protocol will have similar efficacy to the original treatment protocol and will be as well or better received by participants. We hypothesize that the intervention will be shown to be efficacious for improving pain and pain-related concerns among members of this population and that the treatment will be well received by participants.

DETAILED DESCRIPTION:
This study is being conducted to examine the efficacy of a revised version of an online chronic pain intervention tailored specifically for military, RCMP, and veterans. The original intervention is an online psychotherapy for chronic pain that was developed using materials derived from cognitive behavioural therapy (CBT) and acceptance and commitment therapy (ACT) and has thus been described as an acceptance-based behavioural therapy (ABBT). For the purposes of this study, the revised intervention is known as ABBT-R. The revised protocol was developed based on feedback from participants who had engaged with the original version and who participated in a focus group study about their experiences. It is hoped that the revised treatment protocol will have similar efficacy to the original treatment protocol and will be as well or better received by participants. The investigators hypothesize that the intervention will be shown to be efficacious for improving pain and pain-related concerns among members of this population and that the treatment will be well received by participants.

The investigators developed an online psychotherapy for chronic pain that utilizes elements of CBT and ACT, and tailored the content specifically to military and police populations. A pilot study evaluating the efficacy of this 8-week, online, acceptance-based behavioral therapy (ABBT) for chronic pain showed reductions in fear of movement/re-injury and pain-related catastrophizing and increases in pain acceptance from pre- to post-treatment. A randomized controlled trial comparing the same ABBT to a waitlist control condition showed the treatment was efficacious for improving pain acceptance, fear of movement/re-injury, and pain-related disability, with treatment effects ranging from large to very large. A recently conducted focus-group study with individuals who had engaged with the treatment provided information about ways to improve the materials to better meet the needs and sensitivities of this population. Based on the feedback from these participants, the original online ABBT has been revised and updated, and the current study will pilot test this new version.

The primary objective of this study is to examine the efficacy of a revised, updated version of an online acceptance-based behavioural therapy (ABBT-R) for addressing chronic pain in military, RCMP, and Veterans of these forces. The secondary objective of this study is to evaluate the impact of the therapy on psychological concerns frequently related to chronic pain in the population to be studied (military, veterans and RCMP/retired RCMP). A tertiary objective of this study is to assess patient satisfaction with the intervention. As revisions to the program were made based on participant feedback, the researchers are interested to know if the modifications made resulted in a more acceptable/satisfying treatment experience.

The study intervention is a revised, updated version of a previously studied eight-module (8-week) online, acceptance-based behavioural therapy (ABBT) for chronic pain that was tailored specifically to a military, RCMP, and veteran population. The revised version of the intervention, known as ABBT-R, is a six-module (6-week) version of the original ABBT. Although outcomes for individuals who completed the original ABBT intervention were favourable, drop-out rates were high. In efforts to improve the treatment to reduce drop-out rates, the investigators conducted a focus group study with previous participants who had completed the program. Participants suggested a reduction to the length of the treatment as many felt the material could be covered in a shorter amount of time. For this reason, the revised version of the program, ABBT-R, has been reduced to six modules to be completed over a period of six weeks, thereby reducing the length of the treatment. No primary content was removed from the program; however, redundancies were removed, and explanations of concepts were simplified and reduced in length where appropriate. As well, content that was deemed either unpleasant or inappropriate for the intended population was revised or removed.

The online treatment material is administered via the WebCAPSI Therapy program, an online password-protected program which allows participants to progress through the modules at their own pace. Each module is designed to cover a component of ABBT and facilitates understanding of the material through audio files, vignettes, text-based material, and homework exercises/assignments. Modules are designed to be completed in 60 minutes or less and participants have the option to return to the program and the modules as often as they like over the course of the intervention. Upon completion of each module, facilitated through the WebCAPSI Therapy program, participants complete an online assignment in which they provide their responses to three randomly selected questions they previously encountered throughout the module. The primary clinician responds to each online assignment through the WebCAPSI Therapy program within 24-hours of its online submission, providing feedback and encouragement.

Based on a recommendation from the HREB during the pilot study of the original ABBT, to incorporate an element of face-to-face contact between participants and the primary clinician during their engagement with the online materials, optional biweekly group sessions are also offered to participants. In the initial optional group session, the clinician provides an overview of the treatment with a specific focus on what to expect in the first two online modules. Each subsequent session revolves around discussion of participant experiences with the previous two online modules, and an overview of what to expect in the next two. Participants who choose not to participate in the group sessions instead participate in individual check-in sessions with the primary clinician at the beginning, mid-point, and end-point of treatment. Throughout their engagement with the intervention, participants can contact the clinician by sending a message through the WebCAPSI Therapy website or by phoning the clinician directly.

The study is a pilot study of an updated and revised version of an existing efficacious therapy. The study uses a single-subject design in which individuals serve as their own controls as a first step in evaluating the efficacy of the revised intervention. The study is an open label, single site, single arm, pilot study. The primary goal of the study is to examine the efficacy of the ABBT-R program via comparison of pre-treatment and post-treatment scores on measures of pain and other related concerns, as well as examination of participant satisfaction with the program. The researchers hypothesize that there will be a reduction in chronic pain symptoms and related concerns following completion of ABBT-R, and that the revised version will be rated as satisfactory by participants.

The source of potential participants is an existing waitlist for chronic pain treatment at the OSI Clinic. Recruitment will proceed via contact by one of the study personnel who has access to the waiting list, as a treatment provider at the clinic. The study personnel will describe the treatment and the study to the potential participants, advise them that they can receive treatment whether they participate in the study or not, and ascertain their willingness to participate.

Potential participants will be told that they are being contacted because they are on the waiting list for chronic pain treatment at the clinic and asked if they are still wishing to receive treatment at the clinic for their chronic pain. Those who indicate they wish to receive treatment will be told about the standard chronic pain treatment at the clinic and advised that the original treatment materials have recently been revised and updated, and that we are doing a research study to determine whether the revised version of the treatment is as effective as the original version.

Participants will be told that if they do not wish to be a part of the study, they have the option of receiving treatment with either the original version or the updated, revised version of the treatment. All individuals wishing to receive treatment will be screened for appropriateness for the treatment, and for those indicating willingness to be a part of the study, the Informed Consent Form will be reviewed with them over the phone and arrangements will be made for a copy of the form to be mailed to them for their signature, with a stamped, return-addressed envelope.

The investigators aim to recruit 34 participants to have adequate power to test the key hypotheses. Statistical analyses will be conducted using SPSS version 27.0. Standard procedures for data screening, preparation, assessing assumptions of normality, and dealing with missing data and outliers will be used prior to hypothesis testing. Reliability for each of the measures used in the study will be calculated using Cronbach's alpha. The primary and secondary hypotheses will be tested using paired sample t-tests to compare participants' pre-, and post-treatment scores on the various measures of chronic pain and other related concerns (i.e., depression, PTSD, and quality of life). The tertiary hypothesis will be examined by comparing participants' scores on the client satisfaction questionnaire to published norms using an independent samples t-test. Effect sizes will be calculated for all outcomes.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, individuals must meet all the following criteria:

  1. Be either an actively serving or Veteran member of the Canadian Armed Forces or Royal Canadian Mounted Police
  2. Be over the age of 18
  3. Have been referred to the Winnipeg Operational Stress Injury Clinic for treatment
  4. Report chronic pain of duration six months or longer
  5. Report that they are seeking treatment for their chronic pain
  6. Have access to a computer at least once per week for a 60-minute duration
  7. Agree to receive the revised/updated version of the clinic's standard chronic pain treatment
  8. Provide a signed and dated informed consent form

Exclusion Criteria:

* An individual who meets any of the following criteria at baseline will be excluded from participation in this study:

  1. Current uncontrolled or untreated psychosis
  2. Significant suicide risk
  3. Seriously impaired concentration
  4. Significant cognitive impairment
  5. Unstable living situation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain ratings | From pre-treatment to post-treatment (approximately 6 weeks)
  Changes are expected on the McGill Pain Questionnaire-Short Form. On this measure, a higher score means a worse outcome. The primary scale will be examined, which has a minimum of 0 and maximum of 45.
Change in pain-related disability | From pre-treatment to post-treatment (approximately 6 weeks)
  Changes are expected on the Pain Disability Index. On this measure, a higher score means a worse outcome. The minimum score is 0 and the maximum is 70.
Change in pain-related catastrophizing | From pre-treatment to post-treatment (approximately 6 weeks)
  Changes are expected on the Pain Catastrophizing Scale. On this measure, a higher score means a worse outcome. The minimum score is 0 and the maximum is 52.
Change in pain-related acceptance | From pre-treatment to post-treatment (approximately 6 weeks)
  Changes are expected on the Chronic Pain Acceptance Questionnaire-Revised. On this measure, a higher score means a better outcome. The minimum score is 20 and the maximum is 120.
Change in pain-related fear of movement | From pre-treatment to post-treatment (approximately 6 weeks)
  Changes are expected on the Tampa Scale of Kinesiophobia- 11 item version. On this measure, a higher score means a worse outcome. The minimum score is 11 and the maximum is 44.

SECONDARY OUTCOMES:
Change in depression symptoms | From pre-treatment to post-treatment (approximately 6 weeks)
  Changes are expected on the Patient Health Questionnaire-9. On this measure, a higher score means a worse outcome. The minimum score is 0 and the maximum is 27.
Change in posttraumatic stress symptoms | From pre-treatment to post-treatment (approximately 6 weeks)
  Changes are expected on the Posttraumatic Checklist - DSM5 version. On this measure, a higher score means a worse outcome. The minimum score is 0 and the maximum score is 80.
Change in overall quality of life | From pre-treatment to post-treatment (approximately 6 weeks)
  Changes are expected on the Short-Form Health Survey - 20 item version. On this measure, a higher score means a better outcome. The minimum score is 20 and the maximum is 91.

OTHER OUTCOMES:
Client satisfaction | End of treatment measure only (at the end of the 6 week trial)
  Client satisfaction will be measured with the Client Satisfaction Questionnaire (CSQ-8) and compared to outcomes from a trial of a previous version of this treatment. The measure has 8 items. Higher scores are associated with better outcomes. The minimum is 8 and the maximum is 32.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Akerblom S, Perrin S, Rivano Fischer M, McCracken LM. The Relationship Between Posttraumatic Stress Disorder and Chronic Pain in People Seeking Treatment for Chronic Pain: The Mediating Role of Psychological Flexibility. Clin J Pain. 2018 Jun;34(6):487-496. doi: 10.1097/AJP.0000000000000561. PMID 29016388
- [Result] Andersson G. Internet interventions: Past, present and future. Internet Interv. 2018 Apr 6;12:181-188. doi: 10.1016/j.invent.2018.03.008. eCollection 2018 Jun. PMID 30135782
- [Result] Blaettler LT, Stewart JA, Gubler DA, Egloff N, von Kanel R, Grosse Holtforth M. Alexithymia moderates effects of psychotherapeutic treatment expectations on depression outcome in interdisciplinary chronic pain treatment. J Psychosom Res. 2019 Jul;122:69-72. doi: 10.1016/j.jpsychores.2019.04.010. Epub 2019 Apr 13. PMID 31010581
- [Result] Buhler, J., Holens, P., & Sharpe, D. (2021). A Randomized Controlled Trial of an Online Acceptance and Commitment Therapy-based Intervention for Chronic Pain for Military and Police. Military Behavioral Health. https://doi.org/10.1080/21635781.2021.1982086
- [Result] Buhrman M, Gordh T, Andersson G. Internet interventions for chronic pain including headache: A systematic review. Internet Interv. 2016 Jan 3;4:17-34. doi: 10.1016/j.invent.2015.12.001. eCollection 2016 May. PMID 30135787
- [Result] Fayaz A, Croft P, Langford RM, Donaldson LJ, Jones GT. Prevalence of chronic pain in the UK: a systematic review and meta-analysis of population studies. BMJ Open. 2016 Jun 20;6(6):e010364. doi: 10.1136/bmjopen-2015-010364. PMID 27324708
- [Result] Gaskin DJ, Richard P. The economic costs of pain in the United States. J Pain. 2012 Aug;13(8):715-24. doi: 10.1016/j.jpain.2012.03.009. Epub 2012 May 16. PMID 22607834
- [Result] Gore M, Sadosky A, Stacey BR, Tai KS, Leslie D. The burden of chronic low back pain: clinical comorbidities, treatment patterns, and health care costs in usual care settings. Spine (Phila Pa 1976). 2012 May 15;37(11):E668-77. doi: 10.1097/BRS.0b013e318241e5de. PMID 22146287
- [Result] Holens, P., Buhler, J., & Klassen, K. (2017). Preliminary Trial of an Online Acceptance-Based Behavioural Treatment for Military, Police, and Veterans with Chronic Pain. Journal of Military, Veteran and Family Health (3), 12-21. https://doi.org/10.3138/jmvfh.4315
- [Result] Hunfeld JA, Perquin CW, Duivenvoorden HJ, Hazebroek-Kampschreur AA, Passchier J, van Suijlekom-Smit LW, van der Wouden JC. Chronic pain and its impact on quality of life in adolescents and their families. J Pediatr Psychol. 2001 Apr-May;26(3):145-53. doi: 10.1093/jpepsy/26.3.145. PMID 11259516
- [Result] Kemler MA, Furnee CA. The impact of chronic pain on life in the household. J Pain Symptom Manage. 2002 May;23(5):433-41. doi: 10.1016/s0885-3924(02)00386-x. PMID 12007761
- [Result] Libbrecht, A., Paluszek, M., Romaniuk, A., & Holens, P.L., (2021). A Patient-Informed Qualitative Review of an Online Chronic Pain Treatment for Military, Police, and Veterans. Journal of Military, Veteran, and Family Health. https://doi.org/10.3138/jmvfh-2021-0047
- [Result] Mathias SD, Kuppermann M, Liberman RF, Lipschutz RC, Steege JF. Chronic pelvic pain: prevalence, health-related quality of life, and economic correlates. Obstet Gynecol. 1996 Mar;87(3):321-7. doi: 10.1016/0029-7844(95)00458-0. PMID 8598948
- [Result] Mehta S, Peynenburg VA, Hadjistavropoulos HD. Internet-delivered cognitive behaviour therapy for chronic health conditions: a systematic review and meta-analysis. J Behav Med. 2019 Apr;42(2):169-187. doi: 10.1007/s10865-018-9984-x. Epub 2018 Nov 1. PMID 30387008
- [Result] Rini C, Williams DA, Broderick JE, Keefe FJ. Meeting them where they are: Using the Internet to deliver behavioral medicine interventions for pain. Transl Behav Med. 2012 Mar;2(1):82-92. doi: 10.1007/s13142-011-0107-2. PMID 22924084
- [Result] Rosland AM, Heisler M, Piette JD. The impact of family behaviors and communication patterns on chronic illness outcomes: a systematic review. J Behav Med. 2012 Apr;35(2):221-39. doi: 10.1007/s10865-011-9354-4. Epub 2011 Jun 21. PMID 21691845
- [Result] Schopflocher D, Taenzer P, Jovey R. The prevalence of chronic pain in Canada. Pain Res Manag. 2011 Nov-Dec;16(6):445-50. doi: 10.1155/2011/876306. PMID 22184555
- [Result] Van Den Kerkhof, E. G., Carley, M. E., Hopman, W. M., Ross-White, A., & Harrison, M. B. (2014). Prevalence of chronic pain and related risk factors in military veterans: A systematic review. JBI Database of Systematic Reviews and Implementation Reports, 12(10), 152-186. https://doi:10.11124/jbisrir-2014-1720
- [Result] Vallejo MA, Ortega J, Rivera J, Comeche MI, Vallejo-Slocker L. Internet versus face-to-face group cognitive-behavioral therapy for fibromyalgia: A randomized control trial. J Psychiatr Res. 2015 Sep;68:106-13. doi: 10.1016/j.jpsychires.2015.06.006. Epub 2015 Jun 20. PMID 26228408
- [Result] VanDenKerkhof EG, VanTil L, Thompson JM, Sweet J, Hopman WM, Carley ME, Sudom K. Pain in Canadian Veterans: analysis of data from the Survey on Transition to Civilian Life. Pain Res Manag. 2015 Mar-Apr;20(2):89-95. doi: 10.1155/2015/763768. Epub 2015 Jan 20. PMID 25602711
- [Result] Zanocchi M, Maero B, Nicola E, Martinelli E, Luppino A, Gonella M, Gariglio F, Fissore L, Bardelli B, Obialero R, Molaschi M. Chronic pain in a sample of nursing home residents: prevalence, characteristics, influence on quality of life (QoL). Arch Gerontol Geriatr. 2008 Jul-Aug;47(1):121-8. doi: 10.1016/j.archger.2007.07.003. Epub 2007 Nov 19. PMID 18006088